CLINICAL TRIAL: NCT05475041
Title: Simultaneous Resection of Colorectal Cancer and Synchronous Liver Metastases: What Determines the Risk of Unfavorable Outcomes? A Retrospective International Multicenter Study
Brief Title: Perioperative Outcomes of Simultaneous Colorectal and Liver Resections
Acronym: SIMULT
Status: Completed | Type: Observational
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Collaborators: University of Amsterdam (Other); Universita di Verona (Other); Umberto I Mauriziano Hospital Turin (Unknown); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); IRCCS San Raffaele (Other); University Hospital Padua (Unknown); Riuniti Hospital Polytechnic University of Marche Ancona (Unknown); Clinica Universidad de Navarra Pamplona (Unknown); Groeninge Hospital Kortrijk (Unknown); Oslo University Hospital and Institute of Medicine (Unknown); The Queen Elizabeth Hospital (Other); Antoine Béclère Hospital Paris (Unknown); Moscow Clinical Research Centre (Unknown); University Hospital of Girona Dr. Josep Trueta (Network); University Hospital Southampton NHS Foundation Trust (Other); Università Cattolica del Sacro Cuore-IRCCS Rome (Unknown)
Responsible Party: Sponsor
Other Study IDs: NP5467
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer Metastatic; Surgical Procedure, Unspecified
Keywords: colorectal cancer; synchronous colorectal liver metastases; simultaneous resection; postoperative outcomes
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Minor liver resection: Minor liver resection (<3 contiguous segments) in the anterolateral segments
- Technically major liver resection: Minor liver resection (<3 contiguous segments) in the posterosuperior segments (Segment 1,4a,7,8)
  Interventions: Procedure: Technically major liver resection
- Major liver resection: Major liver resection (3 or more contiguous segments)
  Interventions: Procedure: Major liver resection

INTERVENTIONS:
Procedure: Major liver resection — Major liver resection (3 or more contiguous segments)
  Groups: Major liver resection
Procedure: Technically major liver resection — Minor liver resection (<3 contiguous segments) in the posterosuperior segments (segment 1,4a,7,8)
  Groups: Technically major liver resection

SUMMARY:
The use of a simultaneous resection in patients with synchronous colorectal liver metastases has increased over the past decades. However, it remains unclear when a simultaneous resection is beneficial and when it should be avoided. The objective of this retrospective study is therefore to compare the outcomes of a simultaneous resection for synchronous colorectal liver metastases in different settings, and to assess which factors are independently associated with unfavorable outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Elective minimally invasive or open simultaneous resection of colorectal cancer and synchronous colorectal liver metastases

Exclusion Criteria:

* (Partially) robotic-assisted or thoracoscopic procedures
* First stage of associating liver partition and portal vein ligation for staged hepatectomy (ALPPS)
* Patients that underwent major concurrent procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that underwent an elective minimally invasive or open simultaneous resection of colorectal cancer and synchronous colorectal liver metastases in 17 hepato-biliary referall centers in the time period from January 2004 to December 2019
Sampling Method: Non-Probability Sample
Enrollment: 766 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Major complications | 30 days postoperatively
  Severe complications (Clavien-Dindo grade 3a or higher) related to the surgical procedure

SECONDARY OUTCOMES:
Overall complications | 30 days postoperatively
  Overall complications related to the surgical procedure
Length of hospital stay | 30 days postoperatively
  The length of hospital stay for the surgical procedure
R0 resection margin | 30 days postoperatively
  Proportion of patients in whom a microscopically radical resection of both the primary colorectal carcinoma and the liver metastases was performed.
Intraoperative blood loss | During the surgical procedure
  Intraoperative blood loss in milliliters
Operative time | During the surgical procedure
  Operative time in minutes
Conversion to open surgery | During the surgical procedure
  Intra-operative conversion to an open or hand-assisted procedure in the minimally invasive group
Mortality | 90 days postoperatively
  Postoperative mortality
Red blood cell transfusion | During the surgical procedure
  Intraoperative red blood cell transfusion
Intraoperative incidents | During the surgical procedure
  Intraoperative unfavourable incidents

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The data of this study will be available from the corresponding author, Professor Mohammed Abu Hilal, upon reasonable request. The data are not publicly available since this could compromise the privacy of research participants.

REFERENCES:
- [Derived] Sijberden JP, Zimmitti G, Conci S, Russolillo N, Masetti M, Cipriani F, Lanari J, Gorgec B, Benedetti Cacciaguerra A, Rotellar F, D'Hondt M, Edwin B, Sutcliffe RP, Dagher I, Efanov M, Lopez-Ben S, Primrose JN, Giuliante F, Spinelli A, Chand M, Alvarez S, Langella S, Nicosia S, Ruzzenente A, Vivarelli M, Cillo U, Aldrighetti L, Jovine E, Ferrero A, Guglielmi A, Besselink MG, Abu Hilal M. Simultaneous resection of colorectal cancer and synchronous liver metastases: what determines the risk of unfavorable outcomes? An international multicenter retrospective cohort study. Int J Surg. 2023 Mar 1;109(3):244-254. doi: 10.1097/JS9.0000000000000068. PMID 37093069